CLINICAL TRIAL: NCT01390857
Title: Special Drug Use Investigation for VALTREX (Valaciclovir) (Pediatrics Chickenpox)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112323
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Valacyclovir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric patients prescribed valaciclovir: Pediatric patients with chickenpox prescribed valaciclovir during study period.
  Interventions: Drug: Valaciclovir

INTERVENTIONS:
Drug: Valaciclovir

SUMMARY:
The purpose of this post-marketing surveillance study is to collect and assess information on safety and efficacy of valaciclovir in pediatric patients with chickenpox

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with chickenpox (aged less than 15 years old).

Exclusion Criteria:

* Patients with a history of hypersensitivity to the ingredients of valaciclovir or acyclovir.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Japanese pediatric patients with chickenpox (aged less than 15 years old)
Sampling Method: Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This post-marketing surveillance (PMS) study was designed to evaluate the safety and efficacy of valaciclovir in pediatric participants with chickenpox.
Groups:
- Valaciclovir: VALTREX Caplets: 1000 milligrams (mg) 3 times daily for pediatric participants whose weight is 40 kilograms (kg) or more. VALTREX Granules: 25 mg/kg 3 times daily.
Period: Overall Study
Arm/Group | Valaciclovir
Started | 379
Completed | 369
Not Completed | 10
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 1
Not completed — No Visit after the First Visit | 7

BASELINE CHARACTERISTICS:
Arm/Group | Valaciclovir
Number analyzed (Participants) | 369
Age, Customized [Number; unit: Participants] — The number of participants in the indicated age groups was recorded. Baseline characteristics were collected in members of the Intent-to-Treat Safety Population, comprised of all participants to whom the drug was administered, excluding 10 withdrawal participants.
  Participants
    >=1 month to <1 year | 16
    >=1 to <7 years | 311
    >=7 to <=13 years | 42
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected in members of the Intent-to-Treat Safety Population, comprised of all participants to whom the drug was administered, excluding 10 withdrawal participants.
  Participants
    Female | 156
    Male | 213
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected in members of the Intent-to-Treat Safety Population, comprised of all participants to whom the drug was administered, excluding 10 withdrawal participants.
  participants
    Japanese | 369

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Serious Adverse Event
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or results in prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. For a list of all serious adverse events occurring during the course of the study, please see the table entitled "Serious Adverse Events" in the Adverse Event section of the results record.
Time Frame: 1 month
Population: Intent-to-Treat Safety Population: all participants to whom the drug was administered, excluding 10 withdrawal participants.
Measure: Number; unit: participants
Arm/Group | Valaciclovir
Number analyzed (Participants) | 369
participants | 0

2. Secondary Outcome: Number of Participants With the Indicated Adverse Drug Reactions
Description: An adverse drug reaction (ADR) is an adverse event whose causal relationship to study drug was not ruled out by the reporting physician. An adverse event is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. For a list of all ADRs occurring during the course of the study, please also see the table entitled "Other (non-serious) adverse events" in the Adverse Event section of the results record.
Time Frame: 1 month
Population: ITT Safety Population
Measure: Number; unit: participants
Arm/Group | Valaciclovir
Number analyzed (Participants) | 369
participants
  Urticaria | 2
  Diarrhoea | 1

3. Secondary Outcome: Number of Participants With Any Unexpected Adverse Drug Reactions
Description: An unexpected adverse drug reaction is an adverse event whose casual relationship to the study drug is not ruled out by the reporting physician and also is not listed in a package insert of the drug.
Time Frame: 1 month
Population: ITT Safety Population
Measure: Number; unit: participants
Arm/Group | Valaciclovir
Number analyzed (Participants) | 369
participants | 0

4. Secondary Outcome: Number of Participants Classified as Effective and Not Effective
Description: The course of symptoms was comprehensively assessed by the investigator on a four-category scale (Improved, Unchanged, Worsen, and Unassessable) before and after the initiation of valaciclovir therapy. "Improved" was regarded as "Effective," and "Unchanged" and " Worsen" were regarded as "Not effective." The two participants classifed as "Not effective" were classified as "Unchanged."
Time Frame: 1 month
Population: Efficacy Analysis Set: all participants assessed for efficacy who completed all study visits; 7 participants did not undergo an efficacy evaluation, and 13 participants failed to visit after the first visit.
Measure: Number; unit: participants
Arm/Group | Valaciclovir
Number analyzed (Participants) | 349
participants
  Effective | 347
  Not effective | 2

ADVERSE EVENTS:
Arm/Group | Valaciclovir
Serious Adverse Events (participants affected / at risk) | 0/369
Other Adverse Events (participants affected / at risk) | 7/369
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valaciclovir (N=369)
Urticaria (Skin and subcutaneous tissue disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.